CLINICAL TRIAL: NCT02081157
Title: Use of GalaFlex in Ptotic Breast
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Collaborators: Tepha, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1050
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ptotic Breast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Breast Mastopexy with or without reduction using GalaFlex Mesh: Breast mastopexy with or without reduction, using GalaFLEX mesh
  Interventions: Device: GalaFlex Mesh

INTERVENTIONS:
Device: GalaFlex Mesh

SUMMARY:
This study is to assess the physician preference in the clinical performance of the GalaFLEX mesh in soft tissue reinforcement during elective (cosmetic) plastic surgery to the breast, in particular the breast lift mastopexy and breast reduction procedures

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to understand the risks and benefits of participating in the study and must be willing to sign and date the Informed Consent Form for this study approved by the Institutional Review Board (IRB.)
2. Be at least 21 years of age.
3. Be willing and able to comply with the requirements of the protocol.
4. Be willing to refrain from participating in any other investigational interventional study while enrolled in this study.
5. Female subjects must have a negative pregnancy test within the last 24 hours timeline and have no intentions of becoming pregnant during participation in the study, or be sterilized.

Exclusion Criteria:

1. Subjects unwilling or unable to give written consent to participate in the investigation or unable to comply with the requirements of the protocol.
2. Subjects with known severe allergies manifested by a history of anaphylaxis or allergy to GalaFLEX mesh, poly-4-hydroxybutyrate (P4HB), a resorbable polymer, or silicone.
3. Subjects with known active infection and/or who received or are targeted to receive immunosuppressive therapy over the course of the study (such as rheumatoid arthritis).
4. Subjects who received any experimental drug or device within the previous three months.
5. Female subjects who were pregnant or lactating or were intending to become pregnant during the period of the study, or who would not use an adequate method of contraception (contraceptive pill, intra-uterine device) for the duration of the study.
6. Possessed any psychological condition, or was under treatment for any condition which, in the opinion of the Investigator and/or consulting physicians(s), would constitute an unwarranted risk.
7. Have collagen-vascular, connective disease, or bleeding disorders.
8. Have a BMI that is greater than or equal to 30.
9. Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability.
10. Have an autoimmune disease, an immune deficiency, or is on immune suppression drugs.
11. Currently have an alcohol/substance abuse problem or have had a relapse within 1 year prior to screening visit.
12. Have concomitant unrelated condition of breast/chest wall/skin.
13. Have undergone previous breast surgery with the exception of breast biopsy.
14. Subject is currently a smoker or is a prior smoker who quit in the last 12 months.
15. Currently involved with claims for, or is accepting workers compensation.
16. Currently engaged in medical malpractice litigation.

    -

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with ptotic breasts having elective mastopexy, with or without reduction, with the use of GalaFLEX mesh.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
The primary outcome for study success is defined as ptosis correction and maintenance of the surgical correction | 1year
  Correction of ptosis at 3 months must be Grade 0, Pseudoptosis, or Grade 1, and maintenance of ptosis correction at 12 months is demonstrated by a classification of ptosis Grade 1 or less

OTHER OUTCOMES:
Long term visibility: Mammography and ultrasound will be used to evaluate the presence of the mesh or potential for mesh interference in evaluation of the breast tissue. | 1 year
  Long term visibility
Investigator satisfaction with the surgical implantation/usage of GalaFLEX Scaffold based on a satisfaction questionnaire completed at procedural and follow up timepoints | 1 year
  To determine the role that GalaFLEX scaffold plays in MD's perception of the ability to obtain a successful result, MD's provide assessments of the surgical procedures such as mesh handling, ease of placement. At follow up timepoints, a satisfaction questionnaire is completed to assess satisfaction with overall procedural results
Patient satisfaction based on a survey | 1 year
  Patient satisfaction
Adverse event summary | 1 year
  Adverse Events reported in the study will be evaluated for attribution to the devoce/procedure

CONTACTS AND LOCATIONS:
Overall Officials: Connie Garrison, Study Director — Tepha, Inc.

IPD SHARING:
Plan to Share IPD: No